CLINICAL TRIAL: NCT05382936
Title: A Phase 1, Open-label, Dose-escalation Study of the PI3K Inhibitor SL-901 in Patients With Advanced Solid Tumors
Brief Title: Study of the PI3K Inhibitor SL-901 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped after careful consideration of the landscape of similar drugs and evolving standard of care.
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STML-901-0119
Record Dates: First submitted 2021-10-21; First posted 2022-05-19 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Patients were assigned to the QD or BID regimen based on cohort assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QD Regimen (Experimental): Patients in the QD regimen took study medication once daily.
  Interventions: Drug: SL-901
- BID Regimen (Experimental): Patients in the BID regimen took study medication twice daily.
  Interventions: Drug: SL-901

INTERVENTIONS:
Drug: SL-901 — Patients took study medication daily, with dosage based on their assigned cohort and regimen.

SUMMARY:
Study STML-901-0119 was a dose-escalation study evaluating multiple doses and schedules of orally administered SL-901 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Study STML-901-0119 was a multi-center, open-label, dose-escalation, and regimen-finding study aimed to investigate the safety, pharmacokinetics (PK), and pharmacodynamics of SL-901 in patients with advanced solid tumors. This study initially included two parts: Part 1a, which used a 3+3 dose-escalation design to determine the maximum tolerated dose and an appropriate dosing regimen of SL-901 when administered on both once-daily (QD) and twice-daily (BID) schedules; Part 1b, which was intended to evaluate the clinical activity of SL-901 at the selected dose in patients with advanced solid tumors with specific genetic alterations.

The study was stopped after careful consideration of the landscape of similar drugs and evolving standard of care. As a result, Part 1b was not initiated. In Part 1a, eligible patients were enrolled to receive SL-901 orally on a 28-day cycle. Study enrollment was conducted in 2 centers in the United Kingdom, and patients were assigned to either the QD or BID dosing regimen based on their cohort assignment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older.
2. Population by study stage:

   1. Part 1a: Patients with advanced, metastatic, and/or progressive solid tumors for whom there is no effective standard therapy available.
   2. Part 1b: Patients with histologically confirmed, advanced, metastatic, unresectable, and/or progressive solid tumors for whom there is no effective standard therapy available and their PI3K or DNA-PK pathway is deregulated or their tumor genetic profile has been shown to correlate with sensitivity to PI3K and/or DNA-PK inhibition based on clinical and preclinical experience. Specific criteria will be determined based on ongoing experiments and will be introduced in a future protocol amendment.
3. Evaluable or measurable disease.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
5. Able to take oral medications.
6. If a woman of childbearing potential (WOCBP), the patient has a negative serum or urine pregnancy test within 1 week before Cycle 1, Day 1 (C1D1). Refer to Section 8.1.3 for further practical information about contraception.
7. The patient (either male or female) agrees to use acceptable contraceptive methods for the duration of time in the study, and to continue to use acceptable contraceptive methods for 1 month after the last dose of SL-901. Refer to Section 8.1.3 for further practical information about contraception.
8. Able to provide written informed consent.
9. Willing to provide consent for biomarker analysis of existing paraffin-embedded tumor samples.

Exclusion Criteria:

1. Received an investigational anticancer drug within 4 weeks of the first planned SL-901 dose.
2. Received major surgery, radiotherapy, or immunotherapy within 4 weeks of C1D1. Localized palliative radiotherapy is permitted for symptom control.
3. Received chemotherapy regimens with delayed toxicity within 4 weeks (6 weeks for prior nitrosourea or mitomycin C) of C1D1.
4. Received chemotherapy regimens given continuously or on a weekly basis which have limited potential for delayed toxicity within 2 weeks of C1D1.
5. Clinically significant, unresolved toxicity from previous anticancer therapy ≥Grade 2 (except alopecia), as determined by the Investigator using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
6. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
7. Left ventricular ejection fraction <50%.
8. Corrected QT interval (based on Fridericia's formula) >450 msec.
9. Type 1 or 2 diabetes mellitus requiring medication. (In Part 1b, patients with type 2 diabetes mellitus controlled by medication, as indicated by a glycated hemoglobin of ≤7.5% are eligible.)
10. Known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
11. Ongoing systemic bacterial, fungal, or viral infection.
12. History of interstitial pneumonitis.
13. Absolute neutrophil count (ANC) 1.5×10⁹/L.
14. Hemoglobin <10 g/dL.
15. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5x the upper limit of normal (ULN).
16. Known hypersensitivity or allergy to the active ingredient or excipients of SL-901.
17. Breast-feeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Marsden Hospital, Sutton, Surrey
  - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn C. An evaluation of phase I cancer clinical trial designs. Stat Med. 1998 Jul 30;17(14):1537-49. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-f. PMID 9699228
- [Background] Courtney KD, Corcoran RB, Engelman JA. The PI3K pathway as drug target in human cancer. J Clin Oncol. 2010 Feb 20;28(6):1075-83. doi: 10.1200/JCO.2009.25.3641. Epub 2010 Jan 19. PMID 20085938
- [Background] Gatsonis C, Greenhouse JB. Bayesian methods for phase I clinical trials. Stat Med. 1992 Jul;11(10):1377-89. doi: 10.1002/sim.4780111011. PMID 1518998
- [Background] Greenwell IB, Ip A, Cohen JB. PI3K Inhibitors: Understanding Toxicity Mechanisms and Management. Oncology (Williston Park). 2017 Nov 15;31(11):821-8. PMID 29179250
- [Background] Krause G, Hassenruck F, Hallek M. Copanlisib for treatment of B-cell malignancies: the development of a PI3K inhibitor with considerable differences to idelalisib. Drug Des Devel Ther. 2018 Aug 21;12:2577-2590. doi: 10.2147/DDDT.S142406. eCollection 2018. PMID 30174412
- [Background] Liu P, Cheng H, Roberts TM, Zhao JJ. Targeting the phosphoinositide 3-kinase pathway in cancer. Nat Rev Drug Discov. 2009 Aug;8(8):627-44. doi: 10.1038/nrd2926. PMID 19644473
- [Background] Storer BE. Design and analysis of phase I clinical trials. Biometrics. 1989 Sep;45(3):925-37. PMID 2790129

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: SL-901 20 mg: Subjects received SL-901 20 mg for a 28-day treatment cycle at once daily dosing.
- Cohort 2: SL-901 40 mg: Subjects received SL-901 40 mg for a 28-day treatment cycle at both once-daily and twice-daily dosing.
- Cohort 3: SL-901 60 mg: Subjects received SL-901 60 mg for a 28-day treatment cycle at once-daily dosing.
- Cohort 4: SL-901 80 mg: Subjects received SL-901 80 mg for a 28-day treatment cycle at both once-daily and twice-daily dosing.
Period: Overall Study
Arm/Group | Cohort 1: SL-901 20 mg | Cohort 2: SL-901 40 mg | Cohort 3: SL-901 60 mg | Cohort 4: SL-901 80 mg
Started | 3 | 7 | 4 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 4 | 6
Not completed — Progressive Disease | 3 | 5 | 2 | 5
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Deteriorated Performance Status. Unlikely Benefit | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SL-901 20 mg | Cohort 2: SL-901 40 mg | Cohort 3: SL-901 60 mg | Cohort 4: SL-901 80 mg | Total
Number analyzed (Participants) | 3 | 7 | 4 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (10.69) | 54.3 (6.58) | 51.0 (7.75) | 59.5 (14.35) | 54.8 (0.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 1 | 10
  Male | 0 | 4 | 1 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 4 | 5 | 18
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 2 | 5 | 3 | 4 | 14
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: To Identify the MTD, Appropriate Dosing Regimen, PK Profile, and Perform Initial Assessment of the Safety Profile of SL-901
Description: * Safety endpoints include identification of DLTs; rate of TEAEs and SAEs; identification of abnormalities in physical examination, vital signs, clinical laboratory evaluations, and ECG findings.
  * PK endpoints include assessment of SL-901 plasma concentration over time; assessment of any changes in the PK properties of SL-901 between initial administration and steady-state and between cycles of treatment; explore the correlation between PK parameters and toxicity.
Time Frame: Approximately 2 years
Population: Safety Population
Measure: Number; unit: adverse event
Arm/Group | Cohort 1: SL-901 20 mg | Cohort 2: SL-901 40 mg | Cohort 3: SL-901 60 mg | Cohort 4: SL-901 80 mg
Number analyzed (Participants) | 3 | 7 | 4 | 6
adverse event
  Any TEAE | 3 | 7 | 4 | 5
  Any SAE | 1 | 3 | 6 | 0

2. Secondary Outcome: Assess Preliminary Clinical Activity of SL-901 - Best Overall Response
Description: Clinical activity endpoints include the rate of objective response, rate of CR, DOR, PFS, and OS.
Time Frame: Approximately 2 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SL-901 20 mg | Cohort 2: SL-901 40 mg | Cohort 3: SL-901 60 mg | Cohort 4: SL-901 80 mg
Number analyzed (Participants) | 3 | 7 | 4 | 6
Participants
  Best Overall Response - Missing | 0 | 1 | 1 | 0
  Best Overall Response - Stable Disease | 0 | 2 | 1 | 2
  Best Overall Response - Progressive Disease | 3 | 4 | 1 | 4
  Best Overall Response - Not Evaluable | 0 | 0 | 1 | 0

3. Secondary Outcome: Assess Preliminary Clinical Activity of SL-901 - PFS
Description: Progression-free Survival - Investigator's Assessment
Time Frame: Approximately 2 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SL-901 20 mg | Cohort 2: SL-901 40 mg | Cohort 3: SL-901 60 mg | Cohort 4: SL-901 80 mg
Number analyzed (Participants) | 3 | 7 | 4 | 6
Participants
  Subjects with event | 3 | 7 | 2 | 5
  Progressive Disease | 3 | 6 | 2 | 5
  Death | 0 | 1 | 2 | 2
  Censored subjects | 0 | 0 | 2 | 1
  No progressive disease and no death | 0 | 0 | 1 | 1
  No post-baseline and no death | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: All serious and non-SAEs recorded in the study's clinical database from the day of first exposure to SL-901 through 30 days after the last dose of SL-901 (approximately 2 years).
Arm/Group | Cohort 1: SL-901 20 mg | Cohort 2: SL-901 40 mg | Cohort 3: SL-901 60 mg | Cohort 4: SL-901 80 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/7 | 2/4 | 2/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/7 | 3/4 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 4/4 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SL-901 20 mg (N=3) | Cohort 2: SL-901 40 mg (N=7) | Cohort 3: SL-901 60 mg (N=4) | Cohort 4: SL-901 80 mg (N=6)
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SL-901 20 mg (N=3) | Cohort 2: SL-901 40 mg (N=7) | Cohort 3: SL-901 60 mg (N=4) | Cohort 4: SL-901 80 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 4 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was stopped after careful consideration of the landscape of similar drugs and evolving standard of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Stemline shall have the right to publish the results of the study
* This is a multi-site study; therefore, publication of results from all sites is expected
* Institution's (PI's) results may be submitted for publication only after multicenter results have been published, 18 months after study completion.
* PI to submit copy of publication/presentation to Stemline for review/comment at least 60 days prior to submission for publication

DOCUMENTS (2):
  • Study Protocol (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT05382936/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT05382936/SAP_001.pdf